CLINICAL TRIAL: NCT03456167
Title: Mobile App Postoperative Home Monitoring After Enhanced Recovery Oncologic Surgery
Acronym: ERAS-OncoRe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health Services, Calgary (Other)
Collaborators: Alberta Cancer Foundation (Other)
Responsible Party: Principal Investigator, Claire Temple-Oberle, Professor, Departments of Surgery and Oncology, Alberta Health Services, Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TomBakerCC
Record Dates: First submitted 2017-12-04; First posted 2018-03-07 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Gynecologic Cancer
Keywords: telemedicine; mobile applications; ERAS; postoperative care; patient satisfaction; breast reconstruction; gynecologic oncology; mastectomy
MeSH Terms: conditions — Breast Neoplasms; Patient Satisfaction | interventions — Aftercare

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile app for follow-up care (Experimental): Participants will use an app to submit photos of their surgical site, QoR15 scores, and EORTC selected adverse events scores daily for 2 weeks post-op & weekly for another 4 weeks. Surgeons will use a wireless interface to access that data and monitor the patient's condition. Participants will complete questionnaires and keep diaries related to satisfaction, medical system encounters, surgical complications, followup-related financial costs, and telemedicine satisfaction at 2 & 6 weeks post-op. They will attend prescribed follow-up appointments with their surgeon with the option to skip 1 or more follow-up appointments dependent on their recovery trajectory & surgeon.
  Interventions: Other: RecoverWell mobile app for follow-up care
- Conventional inperson followup care (No Intervention): The conventional follow-up care group will keep to conventional follow-up schedules of all surgeons involved. They will complete questionnaires and keep diaries related to satisfaction, medical system encounters, surgical complications, and followup-related financial costs at 2 & 6 weeks post-op and attend all scheduled follow up appointments.

INTERVENTIONS:
Other: RecoverWell mobile app for follow-up care — The mobile app follow-up care is an application that can be loaded onto a smartphone. It allows the patient to submit photos of their surgical site, QoR15 scores, and EORTC selected adverse events scores. The information collected is transmitted to members of the surgical team (i.e. the primary surgeon) and used to monitor recovery over the first 6 weeks following surgery.
  Other Names: QoC Health Inc. mobile application; RecoverWell
  Arms: Mobile app for follow-up care

SUMMARY:
This study will assess whether the implementation of a combination of ERAS (Enhanced Recovery After Surgery) protocols and postoperative followup via a smartphone app can offer 1) improved patient satisfaction, 2) virtual patient monitoring without an increase in postoperative emergency room visits, number and severity of postoperative complications, and readmissions, 3) decreased healthcare system costs, and 4) improved patient convenience and reduced patient financial costs. The study will be conducted among women having mastectomy, breast reconstruction, and gynecological oncology procedures. Half of the participants will be assigned to physician monitoring via a smartphone app and half will receive conventional care.

DETAILED DESCRIPTION:
ERAS® (Enhanced Recovery After Surgery) protocols are evidence-based best practices bundled together to revolutionize pre-, intra-, and postoperative care resulting in better patient outcomes, increased patient postoperative satisfaction, and decreased healthcare costs. ERAS® protocols in breast reconstruction and gynecologic oncology have been developed by surgeons from the Tom Baker Cancer Centre and have the sanction of the international ERAS® Society for implementation globally.

As of 2015, the majority of Canadians owned a cell phone. Technological advances in these forms of communications have been shown to positively impact patient experience and reduce healthcare system burdens. Telemedicine delivered healthcare via smartphone apps now include platforms for encouraging healthy behaviors, monitoring chronic healthcare conditions, organizing personal healthcare records, and monitoring postsurgical wounds.

The proposed study would marry these two advances, ERAS® protocols and smartphone technology, to consider how the combination of these two approaches to postsurgical care might enhance patient satisfaction and convenience and minimize financial burden while providing high quality care and monitoring. Additionally, the combination of these approaches has the potential to benefit the healthcare system in a number of ways. By lessening surgery-related length of stay and reducing the number of postsurgical visits, an opportunity for cost-savings is evident. In addition, in a system that is troubled by long wait-times for some procedures, reducing lengths of stay and surgeons' postoperative clinical burden means more patients can be seen and treated in a timely fashion. This is a win-win for the healthcare system and patients. It provides structure for more efficiently caring for post-operative patients in a patient first manner that supports physicians, transforms care, and engages in responsible stewardship of healthcare resources according to the Foundational Strategies developed by Alberta Health Services.

The current study would assess the patient, physician, and healthcare system impact of combining ERAS® protocol-guided oncological surgery with postsurgical patient monitoring via a smartphone app that would lessen patients' postoperative burden when postoperative recovery is uneventful and would alert physicians earlier when things are not going well.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age undergoing breast reconstruction, mastectomy alone, and major gynecologic oncology procedures under ERAS protocols.
* Must own an Android or iOS smartphone, be familiar with basic smartphone technology, be willing to install the app on their phone, to have their phone doubly-encrypted, and to learn the app and camera features of the phone as needed for the study.
* Fluency in English

Exclusion Criteria:

* Lack of fluency in English
* Lack of daily access to a smartphone where the app can be installed and operated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Questionnaire (PSQ-III) - Select Subscales | 6 weeks
  The PSQ-III is a validated questionnaire made up of several subscales and employing a "statement of opinion" response model of 5 response categories (strongly agree, agree, uncertain, disagree, strongly disagree). The subscales being employed in the current study include general satisfaction, communication with your doctor, time spent with doctor, financial aspects, and access/availability/convenience.
Quality of Recovery 15 | 6 weeks
  The Quality of Recovery 15 scale captures patient reported postoperative assessment of various dimensions of health including patient support, comfort, emotions, physical independence, and pain. Patients rate each of the 15 statements from 1 (never) to 10 (always).

SECONDARY OUTCOMES:
Patient-borne Financial Costs of Followup Appointments | 6 weeks
  The costs related to attending one or more surgical followup appointments will be tracked. Participants will maintain a log of all associated expenses.
Total Number of Contacts with Medical System Postoperatively | 6 weeks
  The total number of contacts with the healthcare system postoperatively will be tracked.
Postoperative Complications | 6 weeks
  All complications occurring within the study period will be tracked. This information will be gathered.
Adverse events NCI Version 3 / EORTC | 6 weeks
  Select adverse events including diarrhea, constipation, fever, urinary frequency/urgency, vaginal bleeding, wound complications, and fatigue will be tracked.
Healthcare Professionals' Contact with Study Patients | 6 weeks
  The participating surgeons and study nurses will keep diaries of time spent on patient followup, including followup appointments, receiving and returning phone calls, and tame spent related to virtual monitoring via the smartphone app.
Healthcare Professional Response to Virtual versus Traditional FollowUp Care | 6 weeks
  A telephone interview will be conducted with study surgeons and nursing staff at the end of the study to inquire into the impact on medical professionals conducting conventional versus virtual monitoring of postoperative patients.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Temple-Oberle, MD MSc FRCSC, Principal Investigator — University of Calgary
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for pre- and intra-operative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part I. Gynecol Oncol. 2016 Feb;140(2):313-22. doi: 10.1016/j.ygyno.2015.11.015. Epub 2015 Nov 18. No abstract available. PMID 26603969
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for postoperative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part II. Gynecol Oncol. 2016 Feb;140(2):323-32. doi: 10.1016/j.ygyno.2015.12.019. Epub 2016 Jan 3. No abstract available. PMID 26757238
- [Background] Temple-Oberle C, Shea-Budgell MA, Tan M, Semple JL, Schrag C, Barreto M, Blondeel P, Hamming J, Dayan J, Ljungqvist O; ERAS Society. Consensus Review of Optimal Perioperative Care in Breast Reconstruction: Enhanced Recovery after Surgery (ERAS) Society Recommendations. Plast Reconstr Surg. 2017 May;139(5):1056e-1071e. doi: 10.1097/PRS.0000000000003242. PMID 28445352
- [Background] Armstrong KA, Coyte PC, Brown M, Beber B, Semple JL. Effect of Home Monitoring via Mobile App on the Number of In-Person Visits Following Ambulatory Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 Jul 1;152(7):622-627. doi: 10.1001/jamasurg.2017.0111. PMID 28329223
- [Derived] Temple-Oberle C, Yakaback S, Webb C, Assadzadeh GE, Nelson G. Effect of Smartphone App Postoperative Home Monitoring After Oncologic Surgery on Quality of Recovery: A Randomized Clinical Trial. JAMA Surg. 2023 Jul 1;158(7):693-699. doi: 10.1001/jamasurg.2023.0616. PMID 37043216

DOCUMENTS (1):
  • Informed Consent Form (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT03456167/ICF_000.pdf